CLINICAL TRIAL: NCT00222430
Title: Fluoroscopy Guided Femoral Arterial Access and the Use of Closure Devices: A Randomized Controlled Trial.
Brief Title: Fluoroscopy Guided Femoral Arterial Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11854
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Vascular Access
Keywords: Fluoroscopy; Femoral Artery; Arterial Vascular Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Usual standard coronary angiographic procedure
  Interventions: Procedure: Active Comparator
- B (Experimental): Fluoroscopy-guided coronary angiography
  Interventions: Procedure: Fluoroscopy

INTERVENTIONS:
Procedure: Fluoroscopy — Use of fluoroscopy during arterial insertion of coronary catheter
  Arms: B
Procedure: Active Comparator — Standard coronary angiography technique; no fluoroscopic assistance
  Arms: A

SUMMARY:
The purpose of this study is to compare the use of fluoroscopic guidance, (a commonly used X-ray technique), with the traditional approach, (where the doctors feel for the strongest pulse), to obtain access to the blood vessel in the groin. These two methods are being compared to assess which is faster, safer and more often allows your physician to use an "arterial closure device," a small suture or plug applied at the end of the angiogram where the needle enters your blood vessel if he/she chooses.

DETAILED DESCRIPTION:
Design: A prospective, randomized, controlled clinical trial to study the effectiveness of applying fluoroscopy guided femoral artery access in the cardiac catheterization lab and its effect on the usage of FDA approved femoral artery closure devices. This trial will randomize patients between fluoroscopy guided femoral artery access or femoral artery access using the usual anatomic landmarks and will then study the difference in the ability to use closure devices on the access site.

Purpose: To establish the safety and efficacy of using fluoroscopic assistance to allow access of the common femoral artery rather than its branches and thus increase the ability to use closure devices.

Enrollment: An approximate enrollment of up to 1000 patients (all patients randomized) who will be undergoing cardiac catheterization and who meet all the eligibility criteria at OUMC and VAMC in Oklahoma City.

Duration: The study will be conducted over approximately one year.

Primary Endpoint: Prediction of ability to use femoral artery closure device based on angiographic data of the femoral artery from fluoroscopy arm versus traditional technique arm.

Secondary Endpoints:

1. Compare the incidence of known major side effects of femoral artery puncture between the two methods of access
2. Compare the time and number of attempts needed to obtain arterial access between the two groups of patients.
3. Compare the ability to puncture the common femoral artery using fluoroscopy vs. anatomical landmarks among different levels of trainees (cardiology fellows) and attending cardiologists.
4. Assess whether fluoroscopic guidance is a superior method to obtain access and thus should be used as a training technique for cardiology fellows.

Analytical Subset: Intention-to-treat sample

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over.
* Patients undergoing elective or urgent left heart cath from the femoral approach.
* Willingness to participate and sign the consent form.

Exclusion Criteria:

* Access from site other than the common femoral artery.
* Creatinine >= 3.0mg/dl.
* Graft in the common femoral artery or other surgeries at that site that might have changed the anatomy of the groin.
* Unable or refusal to sign a consent form.
* Patients from the Department of Corrections.
* Pregnant Women
* Undetectable femoral artery pulse.
* Patients undergoing emergent cardiac catheterization for ST elevation MI or unstable ACS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2005-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Prediction of ability to use femoral artery closure device based on angiographic data of the femoral artery from fluoroscopy arm versus traditional technique arm. | 24 hours

SECONDARY OUTCOMES:
Compare the incidence of known major side effects of femoral artery puncture between the two methods of access | 24 hours
Compare the time and number of attempts needed to obtain arterial access between the two groups of patients. | Intraprocedural
Compare the ability to puncture the common femoral artery using fluoroscopy vs. anatomical landmarks among different levels of trainees (cardiology fellows) and attending cardiologists. | Intraprocedural
Assess whether fluoroscopic guidance is a superior method to obtain access and thus should be used as a training technique for cardiology fellows. | End of study analysis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hennebry, M.D., Principal Investigator — University of Oklahoma; Mazen S Abu-Fadel, M.D., Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Abu-Fadel MS, Sparling JM, Zacharias SJ, Aston CE, Saucedo JF, Schechter E, Hennebry TA. Fluoroscopy vs. traditional guided femoral arterial access and the use of closure devices: a randomized controlled trial. Catheter Cardiovasc Interv. 2009 Oct 1;74(4):533-9. doi: 10.1002/ccd.22174. PMID 19626694